CLINICAL TRIAL: NCT00269256
Title: Stress, Environment, and Genetics in Urban Asthma
Brief Title: Stress, Environment, and Genetics in Urban Children With Asthma
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Rosalind Jo Wright M.D.,M.P.H., Assistant Professor, Brigham and Women's Hospital
Other Study IDs: 1322; R01HL080674 (NIH)
Record Dates: First submitted 2005-12-21; First posted 2005-12-23 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-02

CONDITIONS: Asthma; Lung Diseases
MeSH Terms: conditions — Asthma; Lung Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Maternal DNA Child DNA
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate the multiple mechanisms through which stress, physical environment, and genetic predisposition contribute to asthma in urban children.

DETAILED DESCRIPTION:
BACKGROUND:

The study design builds on the ACCESS Study, a prospective pregnancy cohort study begun in 2003 of a cohort from birth to age four. The present study includes two new aims regarding the interaction of stress and genetic or environmental variables, reflecting a more comprehensive conceptualization of the multiple mechanisms by which stress can contribute to asthma. In addition, the current study proposes to follow the cohort until the age of three.

DESIGN NARRATIVE:

The study examines the role of psychosocial stressors in a systems biology framework considering multiple biologic pathways by which stress can contribute to asthma. The investigators will not only study the independent effect of stress on asthma/wheeze phenotypes in early childhood but also will consider stress as a modifier of physical environmental factors (allergens, cigarette smoking, and diesel-related air pollutants) and genetic predisposition on asthma risk. They will determine the independent effect of maternal stress (both prenatal and postnatal) on early childhood asthma phenotypes. They further hypothesize that multi-life stressors prevalent in disadvantaged populations can cumulatively influence immune system development and airway inflammation in early life, thus making the populations more susceptible to other environmental factors and genetic risk factors explaining, in part, observed asthma disparities associated with SES and race/ethnicity. They will take a multi-level approach, measuring both individual-level stress (negative life events, perceived stress, pregnancy anxiety) and community-level stress [neighborhood disadvantage (e.g., percent of subjects living in poverty, percent unemployed), diminished social capital, and high crime/violence rates]. They will also assess the influence of stress on the infant hormonal stress response and on T-helper cell differentiation as reflected in cytokine profiles and IgE expression (a topic or pro inflammatory phenotype). Additional physical environmental (indoor allergens, diesel-related air pollutants, tobacco smoke) and genetic factors will be assessed given their influence on the immune response and expression of early childhood asthma/wheeze. This interdisciplinary approach is unique because researchers are considering the context in which physical exposures and host susceptibility occur, analyzing their multiplicative joint effects and considering multiple biologic pathways, as such it is consistent with the NIH roadmap objectives.

ELIGIBILITY:
Inclusion criteria:

Mothers aged 18 years or more at time of enrollment and speak English or Spanish.

Exclusion criteria: None

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women and their children followed over first 5 years.
Sampling Method: Non-Probability Sample
Enrollment: 959 (Actual)
Dates: Start 2005-09; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rosalind Wright, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham & Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wright RJ, Fisher K, Chiu YH, Wright RO, Fein R, Cohen S, Coull BA. Disrupted prenatal maternal cortisol, maternal obesity, and childhood wheeze. Insights into prenatal programming. Am J Respir Crit Care Med. 2013 Jun 1;187(11):1186-93. doi: 10.1164/rccm.201208-1530OC. PMID 23590260
- [Background] Chiu YH, Coull BA, Cohen S, Wooley A, Wright RJ. Prenatal and postnatal maternal stress and wheeze in urban children: effect of maternal sensitization. Am J Respir Crit Care Med. 2012 Jul 15;186(2):147-54. doi: 10.1164/rccm.201201-0162OC. Epub 2012 May 10. PMID 22582161
- [Background] Peters JL, Cohen S, Staudenmayer J, Hosen J, Platts-Mills TA, Wright RJ. Prenatal negative life events increases cord blood IgE: interactions with dust mite allergen and maternal atopy. Allergy. 2012 Apr;67(4):545-51. doi: 10.1111/j.1398-9995.2012.02791.x. Epub 2012 Feb 6. PMID 22309645
- [Background] Tse AC, Rich-Edwards JW, Koenen K, Wright RJ. Cumulative stress and maternal prenatal corticotropin-releasing hormone in an urban U.S. cohort. Psychoneuroendocrinology. 2012 Jul;37(7):970-9. doi: 10.1016/j.psyneuen.2011.11.004. Epub 2011 Dec 9. PMID 22154479
- [Background] Sternthal MJ, Coull BA, Chiu YH, Cohen S, Wright RJ. Associations among maternal childhood socioeconomic status, cord blood IgE levels, and repeated wheeze in urban children. J Allergy Clin Immunol. 2011 Aug;128(2):337-45.e1. doi: 10.1016/j.jaci.2011.05.008. Epub 2011 Jun 25. PMID 21704362
- [Result] Chiu YH, Coull BA, Sternthal MJ, Kloog I, Schwartz J, Cohen S, Wright RJ. Effects of prenatal community violence and ambient air pollution on childhood wheeze in an urban population. J Allergy Clin Immunol. 2014 Mar;133(3):713-22.e4. doi: 10.1016/j.jaci.2013.09.023. Epub 2013 Nov 4. PMID 24200349